CLINICAL TRIAL: NCT01287065
Title: A Randomised, Repeat-dose, Placebo-controlled, Double-blind Study to Evaluate and Compare the Efficacy of Fluticasone Furoate/Vilanterol Inhalation Powder, When Administered Either in the Morning or in the Evening, in Male and Female Asthmatic Subjects
Brief Title: A Study in Asthmatic Patients to Determine if There is Any Difference in Dosing With Fluticasone Furoate/Vilanterol Inhalation Powder in the Morning or Evening on Lung Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 114624
Record Dates: First submitted 2011-01-27; First posted 2011-02-01 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Fluticasone furoate; Vilanterol; Efficacy; FEV1; FF/VI Inhalation powder
MeSH Terms: conditions — Asthma | interventions — vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- FF(100mcg)/Vilanterol(25mcg) - AM dosing (Experimental): FF(100mcg)/Vilanterol(25mcg) in the morning (approx 09.00) for 14 days (± 2 days).; placebo in evening (approx 21.00) for 14 days (± 2 days).
  Interventions: Drug: FF(100mcg)/Vilanterol(25mcg) AM; Drug: Placebo PM
- FF(100mcg)/Vilanterol(25mcg) - PM dosing (Experimental): Placebo in morning (approx 09.00) for 14 days (± 2 days); FF(100mcg)/Vilanterol(25mcg) in evening (approx 21.00) for 14 days (± 2 days).
  Interventions: Drug: FF(100mcg)/Vilanterol(25mcg) PM; Drug: Placebo AM
- Placebo (Placebo Comparator): Placebo given in morning (approx 09.00) and in evening (approx (21.00) for 14 days (± 2 days).
  Interventions: Drug: Placebo AM; Drug: Placebo PM

INTERVENTIONS:
Drug: FF(100mcg)/Vilanterol(25mcg) AM — Inhalation powder
  Arms: FF(100mcg)/Vilanterol(25mcg) - AM dosing
Drug: FF(100mcg)/Vilanterol(25mcg) PM — Inhalation powder
  Arms: FF(100mcg)/Vilanterol(25mcg) - PM dosing
Drug: Placebo AM — Inhalation powder
  Arms: FF(100mcg)/Vilanterol(25mcg) - PM dosing; Placebo
Drug: Placebo PM — Inhalation powder
  Arms: FF(100mcg)/Vilanterol(25mcg) - AM dosing; Placebo

SUMMARY:
This study will be a repeat-dose, double-blind, randomized, placebo controlled, three-way crossover study in patients with persistent bronchial asthma to compare the effect of morning (AM) and evening (PM) dosing with fluticasone furoate (FF)/Vilanterol (VI) inhalation powder on lung function. Following screening there will be a run-in period of 14 days. There will be 3 treatment periods; drug at AM, drug at PM and placebo, which will last for 14 days each with a 14-21 day washout period between starting the next. Key assessments include; forced expiratory volume in one second (FEV1), peak expiratory flow (PEF), vital signs, electrocardiograms (ECGs), adverse event (AE) monitoring and laboratory safety tests.

DETAILED DESCRIPTION:
This will be a repeat-dose, double-blind, randomized, placebo controlled, three-way crossover study in patients with persistent bronchial asthma to compare the effect of AM and PM dosing with fluticasone furoate (FF)/Vilanterol (VI) inhalation powder(100/25mcg) on lung function. Twenty-four male and female patients will be enrolled in this study to ensure twenty evaluable subjects. After the screening there will be a run-in period of 14 days prior to first dose. Subjects will be dosed for 14 days (± 2 days) in each of the 3 treatment periods, with serial forced expiratory volume in one second (FEV1) measurements taken over a 24 hour period following the Day 14 PM dose in order to determine FEV1 weighted mean (0-24 hours). Peak expiratory flow (PEF) will also be monitored throughout the study, from the start of the run-in period until the end of the third treatment period. Between treatment periods there will be a washout period of 14-21 days. Safety assessments will include vital signs, electrocardiograms (ECGs), adverse event (AE) monitoring and laboratory safety tests, however, with the exception of AEs these will not constitute study endpoints. The results of the study will provide supporting information to understand the implications of time of day of dosing on the therapeutic response to the FF/VI Inhalation Powder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a documented history of persistent asthma, with the exclusion of other significant pulmonary diseases.
* Male or female between 18 and 70 years of age inclusive
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status prior to study enrollment.
  * Child-bearing potential and agrees to use one of the protocol contraception methods.
* All subjects must be using an inhaled corticosteroid (ICS), with or without a short-acting, beta2-receptor agonist (SABA), for at least 12 weeks prior to screening.
* Subjects with a screening pre-bronchodilator FEV1 ≥ 60% of predicted.
* During the screening visit, subjects must demonstrate the presence of reversible airway disease.
* All subjects must be able to replace all their current asthma treatments with albuterol/salbutamol aerosol inhaler at screening for use as needed for the run-in period and throughout the duration of the study. Subjects must be able to withhold albuterol/salbutamol for at least 6 hours prior to study visits.
* Subjects who are current non-smokers, who have not used any inhaled tobacco products in the 12 month period preceding the screening visit.
* Body weight ≥ 50 kg and Body Mass Index (BMI) within the range 19.0-29.9 kg/m2 (inclusive).
* No evidence of significant abnormality in the 12-lead ECG performed at screening.
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) < 2x Upper limit of normal (ULN); alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Capable of giving written informed consent
* Able to satisfactorily use the novel dry powder inhaler.

Exclusion Criteria:

* A history of life-threatening asthma within the last 5 years.
* Culture-documented or suspected bacterial or viral infection that is not resolved within 4 weeks of screening and led to a change in asthma management or, in the opinion of the Investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Any asthma exacerbation requiring oral corticosteroids within 12 weeks of screening or that resulted in overnight hospitalization requiring additional treatment for asthma within 6 months prior to screening.
* A subject has any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation.
* A subject will not be eligible if he/she has clinical visual evidence of oral candidiasis at screening.
* Pregnant females.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within 30 days prior to the first dosing day in the current study.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Any adverse reaction including immediate or delayed hypersensitivity to any beta 2- agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy.
* History of severe milk protein allergy.
* History of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Subjects who have taken high doses of an ICS within 8 weeks of the screening visit or oral steroids within 12 weeks of the screening visit.
* Subjects who have changed their ICS treatment within the last 4 weeks before screening or can be expected to do so during the study.
* History of regular alcohol consumption within 6 months of the study.
* A positive test for Hepatitis B or Hepatitis C within 3 months of screening.
* A positive breath carbon monoxide (CO) test.
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* No subject is permitted to perform night shift work for 1 week prior to screening until completion of the study treatment periods.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Kempsford RD, Oliver A, Bal J, Tombs L, Quinn D. The efficacy of once-daily fluticasone furoate/vilanterol in asthma is comparable with morning or evening dosing. Respir Med. 2013 Dec;107(12):1873-80. doi: 10.1016/j.rmed.2013.07.002. Epub 2013 Nov 5. PMID 24200619
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114624 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114624 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114624 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114624 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114624 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114624 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114624 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Placebo, FF/VI 100/25 µg AM, FF/VI 100/25 µg PM: Participants received placebo, Fluticasone Furoate (FF)/Vilanterol (VI) 100/25 micrograms (µg) AM, and FF/VI 100/25 µg PM in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments once a day (OD) in the evening from a Dry Powder Inhaler (DPI) for 14 days. Each 14 day treatment period was followed by a 14-21 day washout period.
- Sequence 2: Placebo, FF/VI 100/25 µg PM, FF/VI 100/25 µg AM: Participants received placebo, FF/VI 100/25 µg PM, and FF/VI 100/25 µg AM in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments once a day in the evening from a DPI for 14 days. Each 14 day treatment period was followed by a 14-21 day washout period.
- Sequence 3: FF/VI 100/25 µg AM, FF/VI 100/25 µg PM, Placebo: Participants received FF/VI 100/25 µg AM, FF/VI 100/25 µg PM, and placebo in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments once a day in the evening from a DPI for 14 days. Each 14 day treatment period was followed by a 14-21 day washout period.
- Sequence 4: FF/VI 100/25 µg AM, Placebo, FF/VI 100/25 µg PM: Participants received FF/VI 100/25 µg AM, placebo, and FF/VI 100/25 µg PM in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments once a day in the evening from a DPI for 14 days. Each 14 day treatment period was followed by a 14-21 day washout period.
- Sequence 5: FF/VI 100/25 µg PM, Placebo, FF/VI 100/25 µg AM: Participants received FF/VI 100/25 µg PM, placebo, and FF/VI 100/25 µg AM in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments once a day in the evening from a DPI for 14 days. Each 14 day treatment period was followed by a 14-21 day washout period.
- Sequence 6: FF/VI 100/25 µg PM, FF/VI 100/25 µg AM, Placebo: Participants received FF/VI 100/25 µg PM, FF/VI 100/25 µg AM, and placebo in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments once a day in the evening from a DPI for 14 days. Each 14 day treatment period was followed by a 14-21 day washout period.
Period: Treatment Period 1
Arm/Group | Sequence 1: Placebo, FF/VI 100/25 µg AM, FF/VI 100/25 µg PM | Sequence 2: Placebo, FF/VI 100/25 µg PM, FF/VI 100/25 µg AM | Sequence 3: FF/VI 100/25 µg AM, FF/VI 100/25 µg PM, Placebo | Sequence 4: FF/VI 100/25 µg AM, Placebo, FF/VI 100/25 µg PM | Sequence 5: FF/VI 100/25 µg PM, Placebo, FF/VI 100/25 µg AM | Sequence 6: FF/VI 100/25 µg PM, FF/VI 100/25 µg AM, Placebo
Started | 4 | 4 | 4 | 4 | 5 | 5
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Period: Washout Period 1
Arm/Group | Sequence 1: Placebo, FF/VI 100/25 µg AM, FF/VI 100/25 µg PM | Sequence 2: Placebo, FF/VI 100/25 µg PM, FF/VI 100/25 µg AM | Sequence 3: FF/VI 100/25 µg AM, FF/VI 100/25 µg PM, Placebo | Sequence 4: FF/VI 100/25 µg AM, Placebo, FF/VI 100/25 µg PM | Sequence 5: FF/VI 100/25 µg PM, Placebo, FF/VI 100/25 µg AM | Sequence 6: FF/VI 100/25 µg PM, FF/VI 100/25 µg AM, Placebo
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Sequence 1: Placebo, FF/VI 100/25 µg AM, FF/VI 100/25 µg PM | Sequence 2: Placebo, FF/VI 100/25 µg PM, FF/VI 100/25 µg AM | Sequence 3: FF/VI 100/25 µg AM, FF/VI 100/25 µg PM, Placebo | Sequence 4: FF/VI 100/25 µg AM, Placebo, FF/VI 100/25 µg PM | Sequence 5: FF/VI 100/25 µg PM, Placebo, FF/VI 100/25 µg AM | Sequence 6: FF/VI 100/25 µg PM, FF/VI 100/25 µg AM, Placebo
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Sequence 1: Placebo, FF/VI 100/25 µg AM, FF/VI 100/25 µg PM | Sequence 2: Placebo, FF/VI 100/25 µg PM, FF/VI 100/25 µg AM | Sequence 3: FF/VI 100/25 µg AM, FF/VI 100/25 µg PM, Placebo | Sequence 4: FF/VI 100/25 µg AM, Placebo, FF/VI 100/25 µg PM | Sequence 5: FF/VI 100/25 µg PM, Placebo, FF/VI 100/25 µg AM | Sequence 6: FF/VI 100/25 µg PM, FF/VI 100/25 µg AM, Placebo
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Sequence 1: Placebo, FF/VI 100/25 µg AM, FF/VI 100/25 µg PM | Sequence 2: Placebo, FF/VI 100/25 µg PM, FF/VI 100/25 µg AM | Sequence 3: FF/VI 100/25 µg AM, FF/VI 100/25 µg PM, Placebo | Sequence 4: FF/VI 100/25 µg AM, Placebo, FF/VI 100/25 µg PM | Sequence 5: FF/VI 100/25 µg PM, Placebo, FF/VI 100/25 µg AM | Sequence 6: FF/VI 100/25 µg PM, FF/VI 100/25 µg AM, Placebo
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo, FF/VI 100/25 µg AM, FF/VI 100/25 µg PM in 1 of 6 Seq: All participants received one of the following three treatments in one of three treatment periods from the Dry Powder Inhaler (DPI) for 14 days: placebo in the morning (AM) and evening (PM), Fluticasone Furoate (FF)/Vilanterol (VI) inhalation powder 100/25 micrograms (µg) AM and placebo PM, and FF/VI inhalation powder 100/25 µg PM and placebo AM. Participants were randomized to receive treatment in one of the six following sequences (seq): (1) placebo, FF/VI 100/25 µg AM, FF/VI 100/25 µg PM; (2) placebo, FF/VI 100/25 µg PM, FF/VI 100/25 µg AM; (3) FF/VI 100/25 µg AM, FF/VI 100/25 µg PM, placebo; (4) FF/VI 100/25 µg AM, placebo, FF/VI 100/25 µg PM; (5) FF/VI 100/25 µg PM, placebo, FF/VI 100/25 µg AM; (6) FF/VI 100/25 µg PM, FF/VI 100/25 µg AM, placebo. Each 14 day treatment period was followed by a 14-21 day washout period.
Arm/Group | Placebo, FF/VI 100/25 µg AM, FF/VI 100/25 µg PM in 1 of 6 Seq
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.1 (11.30)
Gender [Count of Participants; unit: Participants]
  Female | 8
  Male | 18
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 25
  Native Hawaiian or other Pacific Islander | 1

OUTCOME MEASURES:

1. Primary Outcome: Weighted Mean Forced Expiratory Volume in One Second (FEV1) Over 0-24 Hours Post-dose on Day 14
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 was measured electronically by spirometry at Day 14. Weighted mean FEV1 was calculated using the Day 14 24-hour serial FEV1 measurements taken at the following time points: pre-dose (Day 14 evening dose), and 3, 6, 9, 12, 15, 18, 21 and 24 hours post-dose (measured in the evening of Day 15). At each time point, the highest of 3 technically acceptable measurements was recorded. The analysis was performed using a mixed effects analysis of covariance model with fixed effect terms for treatment and period; and participant (par.) baseline, period baseline, gender and age fitted as covariates; and par. as a random effect. Par. 122 received FF/VI 100/25 PM in treatment periods 1 and 3 and contributed twice to the summary of FF/VI 100/25 PM (n=25). Par. 123 received Placebo in treatment periods 2 and 3 and contributed twice to the summary of Placebo (n=20).
Time Frame: Pre-dose on Day 14 to 24 hours post-dose
Population: Intent-to-Treat (ITT) Population: all participants who were randomized and received at least one dose of study medication and provided at least one post-dose peak expiratory flow (PEF) or FEV1 measurement. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- Placebo: Participants received placebo in the morning (AM) and evening (PM) from the Dry Powder Inhaler (DPI) for 14 days during one of the three treatment periods. Each 14 day treatment period was followed by a 14-21 day washout period.
- FF/VI 100/25 µg AM: Participants received Fluticasone Furoate (FF)/Vilanterol (VI) inhalation powder 100/25 micrograms (µg) AM and placebo PM from the DPI for 14 days during one of the three treatment periods. Each 14 day treatment period was followed by a 14-21 day washout period.
- FF/VI 100/25 µg PM: Participants received FF/VI inhalation powder 100/25 µg PM and placebo AM from the DPI for 14 days during one of the three treatment periods. Each 14 day treatment period was followed by a 14-21 day washout period.
Arm/Group | Placebo | FF/VI 100/25 µg AM | FF/VI 100/25 µg PM
Number analyzed (Participants) | 20 | 24 | 25
Liters | 2.811 [2.729 to 2.893] | 3.188 [3.112 to 3.265] | 3.233 [3.159 to 3.306]
Statistical Analysis 1: Comparison: Placebo vs FF/VI 100/25 µg AM; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.377, 90% CI 2-sided [0.293 to 0.462] — Mean difference =FF/VI 100/25 µg PM minus Placebo
Statistical Analysis 2: Comparison: Placebo vs FF/VI 100/25 µg PM; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.422, 90% CI 2-sided [0.337 to 0.507] — Mean difference =FF/VI 100/25 µg AM minus Placebo
Statistical Analysis 3: Comparison: FF/VI 100/25 µg AM vs FF/VI 100/25 µg PM; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.044, 90% CI 2-sided [-0.125 to 0.036] — Mean difference =FF/VI 100/25 µg AM minusFF/VI 100/25 µg PM

2. Secondary Outcome: Pre-treatment PEF (AM and PM) on Days 1-12.
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants daily in the morning and evening just prior to each dose, using an electronic peak flow meter, throughout the 14-day Treatment Period. Only the averaged daily AM and PM PEF over Days 2 to 12 was analyzed. The analysis was performed using a mixed effect analysis of covariance model with fixed effect terms for treatment and period; baseline PEF AM and PM, gender and age fitted as covariates; and participant as a random effect. Participant 122 received FF/VI 100/25 PM in treatment periods 1 and 3 and contributed twice to the summary of FF/VI 100/25 PM (n=26). Participant 123 received Placebo in treatment periods 2 and 3 and contributed twice to the summary of Placebo (n=24).
Time Frame: From Day 2 up to Day 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters per minute
Arm/Group | Placebo | FF/VI 100/25 µg AM | FF/VI 100/25 µg PM
Number analyzed (Participants) | 24 | 24 | 26
Liters per minute
  AM Mean PEF, n= 24, 24, 25 | 466.3 [448.8 to 483.9] | 510.4 [492.9 to 527.8] | 535.3 [518.1 to 552.5]
  PM Mean PEF , n= 24, 24, 26 | 453.2 [438.5 to 467.9] | 517.6 [503.0 to 532.2] | 521.4 [507.1 to 535.7]

3. Secondary Outcome: AM and PM Pre-treatment Trough FEV1 on Day 14
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 was measured electronically by spirometry at Day 14. Trough FEV1 is defined as pre-dose (AM and PM) FEV1 measurement taken on Day 14. The analysis was performed using a mixed effects analysis of covariance model with fixed effect terms for treatment and period; and participant baseline, period baseline, gender and age fitted as covariates; and participant as a random effect. Participant 122 received FF/VI 100/25 PM in treatment periods 1 and 3 and contributed twice to the summary of FF/VI 100/25 PM (n=25). Participant 123 received Placebo in treatment periods 2 and 3 and contributed twice to the summary of Placebo (n=23).
Time Frame: Day 14
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | FF/VI 100/25 µg AM | FF/VI 100/25 µg PM
Number analyzed (Participants) | 23 | 24 | 25
Liters
  AM, n=22, 24, 25 | 2.788 [2.684 to 2.892] | 3.191 [3.087 to 3.295] | 3.285 [3.187 to 3.383]
  PM, n=23, 24, 25 | 2.879 [2.775 to 2.982] | 3.153 [3.049 to 3.258] | 3.188 [3.088 to 3.288]

4. Secondary Outcome: Number of Participants With Any Adverse Event (AE) and Any Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, associated with liver injury and impaired liver function defined as alanine aminotransferase >=3 x upper limit of normal (ULN) and total bilirubin >=2 x ULN or international normalised ratio >1.5. Medical or scientific judgment was exercised in deciding whether reporting was appropriate in other situations. Refer to the general AE/SAE module for a list of AEs and SAEs.
Time Frame: From the first dose of the study medication until the Follow-up Visit (up to 18 weeks)
Population: All Subjects Population: all participants who received at least one dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo | FF/VI 100/25 µg AM | FF/VI 100/25 µg PM
Number analyzed (Participants) | 23 | 24 | 25
Participants
  Any AE | 8 | 11 | 12
  Any SAE | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication to the end of the the treatment period (up to Week 18).
Description: SAEs and non-serious AEs were reported for members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of trial medication during the treatment period.
Arm/Group | Placebo | FF/VI 100/25 µg AM | FF/VI 100/25 µg PM
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 8/23 | 11/24 | 12/25
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | FF/VI 100/25 µg AM (N=24) | FF/VI 100/25 µg PM (N=25)
Headache (Nervous system disorders) | 6 | 6 | 8
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 3 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Oral herpes (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.